CLINICAL TRIAL: NCT04823754
Title: Perception of the Doctor/Patient Relationship, Disease and Treatment Among Physicians and Their Patients Treated With Systemic Therapy for Hepatocellular Carcinoma
Brief Title: Perception of the Doctor/Patient Relationship, Disease and Treatment Among Physicians and Their Patients Treated With Systemic Therapy for Hepatocellular Carcinoma "PERCEPTION1"
Acronym: PERCEPTION1
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210481
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma, systemic treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hospitalized patient with advanced hepatocellular carcinoma receiving systemic therapy. — Administation of two surveys to included patients, about the perception of the disease and the expectations related to the treatment.
  The physician will be asked to complete a survey on his or her perception of the prognosis and information received by the patient.

SUMMARY:
atients with cancer face difficult choices that require balancing competing priorities such as survival, functional capacity and symptom relief. Most patients with advanced cancer (>80%) expect their sensitive discussions with physicians about prognosis and treatment choices, in order to be involved in the decision making process. Nevertheless, this kind of discussion is frequently lacking. Consequently, patients often have a biased view of their own prognosis such as an underestimation of disease severity, or unrealistic expectations for cure.

Patients with advanced hepatocellular carcinoma (HCC) may be treated with systemic therapies which may prolong survival, but are not curative. Patients with advanced HCC often report expectations for survival and treatment-related side-effects that differ from their treating physician. Accordingly, communication on prognostic and treatment choices is essential to obtain an accurate understanding of the disease that allows patients to make informed decisions. To the best of our knowledge, a thorough evaluation of the physician-patient communication quality has never been performed in advanced HCC patients.

The aim of our study, is to assess the perception of the expected prognosis, the treatment side-effects; by the patient and by his investigator during the first consultation before the initiation

DETAILED DESCRIPTION:
atients with cancer face difficult choices that require balancing competing priorities such as survival, functional capacity and symptom relief. Most patients with advanced cancer (>80%) expect their sensitive discussions with physicians about prognosis and treatment choices, in order to be involved in the decision making process. Nevertheless, this kind of discussion is frequently lacking. Consequently, patients often have a biased view of their own prognosis such as an underestimation of disease severity, or unrealistic expectations for cure.

Patients with advanced hepatocellular carcinoma (HCC) may be treated with systemic therapies which may prolong survival, but are not curative. Patients with advanced HCC often report expectations for survival and treatment-related side-effects that differ from their treating physician. Accordingly, communication on prognostic and treatment choices is essential to obtain an accurate understanding of the disease that allows patients to make informed decisions. To the best of our knowledge, a thorough evaluation of the physician-patient communication quality has never been performed in advanced HCC patients.

The aim of our study, is to assess the perception of the expected prognosis, the treatment side-effects; by the patient and by his investigator during the first consultation before the initiation

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years of age
2. Patient informed and not objecting to participate in the study
3. Patient with advanced hepatocellular carcinoma.
4. Patient treated with systemic therapy

Exclusion Criteria:

1. Locoregional treatment combined with systemic treatment
2. Pregnancy in progress
3. Candidate for surgery or locoregional therapy
4. Patient with state medical aid (AME)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patient with advanced hepatocellular carcinoma receiving systemic therapy.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the concordance between the patient's perception of his prognosis and treatment side effects with the one of his treating physician. | 12months
  Use of survey completed by the patient and the doctors to assess the primary endpoint

SECONDARY OUTCOMES:
Compare the patient's expectations for the aforementioned items to those of his physician and the degree of concordance between them. | 12 months
  Use of survey completed by the patient and the doctors to assess the primary endpoint
Evaluation of patient satisfaction with the information received during the consultation | 12 months
  Use of survey completed by the patient and the doctors to assess the primary endpoint
Assessment of patient-reported symptoms of anxiety and depression | 12 months
  Use of survey completed by the patient and the doctors to assess the primary endpoint
Evaluate the association between individual prognosis expectation (patient and physician) and data from the available literature. | 12 months
  Use of survey completed by the patient and the doctors to assess the primary endpoint

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Avicenne, Bobigny
  - Assistance Publique - Hôpitaux de Paris, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Loh KP, Mohile SG, Lund JL, Epstein R, Lei L, Culakova E, McHugh C, Wells M, Gilmore N, Mohamed MR, Kamen C, Aarne V, Conlin A, Bearden J 3rd, Onitilo A, Wittink M, Dale W, Hurria A, Duberstein P. Beliefs About Advanced Cancer Curability in Older Patients, Their Caregivers, and Oncologists. Oncologist. 2019 Jun;24(6):e292-e302. doi: 10.1634/theoncologist.2018-0890. Epub 2019 Apr 23. PMID 31015317
- [Background] Yennurajalingam S, Rodrigues LF, Shamieh O, Tricou C, Filbet M, Naing K, Ramaswamy A, Perez-Cruz PE, Bautista MJS, Bunge S, Muckaden MA, Sewram V, Fakrooden S, Noguera-Tejedor A, Rao SS, Liu D, Park M, Williams JL, Lu Z, Cantu H, Hui D, Reddy SK, Bruera E. Perception of Curability Among Advanced Cancer Patients: An International Collaborative Study. Oncologist. 2018 Apr;23(4):501-506. doi: 10.1634/theoncologist.2017-0264. Epub 2017 Nov 20. PMID 29158371
- [Derived] Nault JC, Sritharan N, Verset G, Borbath I, Lequoy M, Allaire M, Regnault H, Colle I, Orlent H, Sinapi I, Moreno C, Larrey E, Sidali S, Hollande C, Amaddeo G, Pol S, Nahon P, Ganne-Carrie N, Levy V, Bloch-Queyrat C; Paris Liver Cancer Group; Trepo E, Bouattour M. Patient and physician expectations regarding disease and treatment of advanced HCC: The prospective PERCEPTION1 study. JHEP Rep. 2024 Aug 22;6(11):101192. doi: 10.1016/j.jhepr.2024.101192. eCollection 2024 Nov. PMID 39741695
- See also: Related Info — http://linkinghub.elsevier.com/retrieve/pii/S0168827818302150